CLINICAL TRIAL: NCT02910492
Title: A Single-Center, Open-Label Exploratory Study of a Novel Laser for Skin Rejuvenation
Brief Title: Study of a Novel Laser for Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-16-EN12
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational Enlighten Device (Experimental): Laser treatment for facial skin rejuvenation with the experimental enLighten Laser
  Interventions: Device: enLighten Laser

INTERVENTIONS:
Device: enLighten Laser — Dual-pulse duration laser for the treatment of skin rejuvenation

SUMMARY:
Single-center study to evaluate the safety and efficacy of an investigational version of the enlighten™ 670nm laser for photo-rejuvenation.

DETAILED DESCRIPTION:
A single-center prospective, open-label uncontrolled exploratory study to evaluate the safety and efficacy of an investigational version of the enlighten™ 670nm laser for photo-rejuvenation.

Subjects will receive laser treatments, and will be followed at 12 weeks post-final treatment. In addition, after each treatment, subjects will complete a 3 day post treatment phone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 18 to 75 years of age (inclusive).
* Fitzpatrick Skin Type I - VI.
* Desires photo-rejuvenation of the skin or improvement in the appearance of acne scarring.
* Subject has visible signs of acne scarring or moderate sun-damaged and/or aging skin in the treatment area with visible areas acne lesions and scars, fine rhytides, lentigines or pigmentation, diffused redness erythema and skin texture
* Subject must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Willing to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treatment area every day for the duration of the study, including the follow-up period.
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s), including injectable agents, for skin rejuvenation during the study and has no intention of having such procedures performed during the course of the study.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant.

Exclusion Criteria:

* Participation in a clinical trial of another drug, or device administered to the target area, during the study.
* Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as laser or light-based procedures or surgery.
* Prior injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler within 6 months of study participation.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications per investigator's discretion.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of retinoid, such as isotretinoin, as applicable, within 6 months of study participation.
* Topical use of retinoid, such as isotretinoin, as applicable, on the treatment area within 1 month of participation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — Cutera Research Center; Omar Ibrahimi, MD, Principal Investigator — Connecticut Skin Institute
Locations (2):
- United States (2):
  - Cutera Research Clinic, Brisbane, California
  - Connecticut Skin Institute, Stamford, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Enlighten Device
Started | 10
Completed | 4
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Enlighten Device
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Degree of Improvement as Assessed by the Investigator (Physician's Global Assessment of Improvement).
Description: Degree of improvement in the treated area at 12 weeks post-final treatment as assessed by the Investigator (Physician's Global Assessment of Improvement).
  Higher scores indicate better outcomes 4= Very Significant Clearing 3=Significant Clearing 2= Moderate Clearing
  1= Mild Clearing 0= No Clearing
Time Frame: 12 weeks post-final treatment, an average of 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Enlighten Device
Number analyzed (Participants) | 4
score on a scale | 1.7 (1.5)

ADVERSE EVENTS:
Time Frame: 12 weeks post final treatment, up to 6 months
Arm/Group | Investigational Enlighten Device
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Enlighten Device (N=10)
Erythema (Skin and subcutaneous tissue disorders) | 10
Edema (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT02910492/Prot_SAP_000.pdf